CLINICAL TRIAL: NCT06270056
Title: Evaluation of Telemedicine Services to Address Urgent Issues Related to Sexual and Reproductive Rights in Ecuador
Brief Title: Evaluation of Telemedicine Medical Abortion Service in Ecuador
Status: Recruiting | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1058
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: abortion
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- early medication abortion via telemedicine: Medication abortion up to 84 days gestation using misoprostol alone regimen consisting of three doses 800mcg (4 tablets of 200mcg misoprostol each) taken every 3 hours. An extra dose (800mcg) may also be taken if there was no bleeding after administering the earlier doses.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Self-administered misoprostol by clients obtaining medication abortion via telemedicine
  Other Names: Cytotec

SUMMARY:
This research seeks to demonstrate that a telemedicine model for the provision of legal abortion services in Ecuador is safe, feasible and acceptable to users requesting a medication abortion and who are less than 12 weeks pregnant.

DETAILED DESCRIPTION:
The purpose of this observational study is to pilot and evaluate the remote provision of medication abortion as part of a telemedicine service that promotes the sexual and reproductive rights of Ecuadorian women. The study aims to enroll 100 participants who contact private sector providers in Ecuador to obtain a medication abortion.

The telemedicine service will be designed to incorporate the standard steps in an in-person medical abortion procedure to ensure that the quality of care provided to each participant is equal to that which one would otherwise receive during visits to a clinic.

Specific objectives include:

* Document interest in the telemedicine model among users who wish to receive a medication abortion with private study providers.
* Document the benefits and disadvantages of the remote care approach perceived by users and providers.
* Document compliance with the requirements established for the provision of telemedicine service for medication abortion within the context of this study.
* Document any obstacles encountered in meeting the requirements of the telemedicine protocol.

Initial-contact and screening for eligibility: Women who contact the study clinic to request a medical abortion and who meet the basic eligibility criteria to terminate their pregnancy using the remote approach will be informed that the study provider offers such an option as part of an investigation. Individuals who express interest in the telemedicine service and are determined as likely to be eligible will have a "TelEvaluation" set up with the study provider, who will give standard pre-abortion counseling (via telephone, video conferencing, etc) and explain the study procedures and process of obtaining informed consent for the study.

TelEvaluation and Informed Consent: During the remote consultation, the provider will explain to the woman what the study consists of and its investigative nature, the benefits and risks of participating in it, all the procedures required, the existing options if she decides not to be enrolled and that she has the right to refuse to participate or leave the study without affecting the medical care she could receive. The consent form will be sent to the woman by email or telephone. If the woman wishes to participate, both she and the provider will sign the form electronically, or obtain her verbal consent, in an application designed for that purpose. Demographic and medical information will be recorded during the TelEvaluation. If required, the provider will assist the client to identify facilities nearby to obtain any tests and have the results sent to the study clinic. No information obtained during or after the TelEvaluation will be sent or included in the study database if informed consent is not obtained.

The study provider will review the test results and information collected at the initial contact and remote consultation (TelEvaluation) and, if available, the ultrasound to determine if the woman is considered eligible to receive telemedicine as part of the study in accordance with the eligibility criteria.

Shipment of study package: Once the study provider confirms the participant's eligibility, the study package will be sent to the participant by certified parcel or other delivery option available in their locality: The package will contain the following:

* 12 misoprostol tablets of 200 mcg each^

  ^The regimen to be used in this study consists of a minimum of three doses (800mcg, i.e. 4 tablets of 200mcg misoprostol each) administered sublingually every three hours. This regimen is supported in the World Health Organization's guidelines.
* 4 additional misoprostol tablets of 200 mcg each, to be used as needed
* Ibuprofen 800 mg (8 tablets)
* Study instruction sheet that includes written instructions on how to use the medications, expected symptoms and side effects, the follow up plan, and what to do in case of an emergency.

Antibiotics, antiemetics and other medications will be prescribed at the discretion of the provider and included with the packet that is shipped. The study provider will provide the participant with the package tracking number. She will be asked to notify the study staff when she receives the package.

Administration of medications: The participant will be instructed to take the first dose of misoprostol on the day she receives the package, provided her gestational age is not more than 84 days. She should take all three doses of misoprostol according to the standard indications for a medical abortion established by the study center. If she does not have bleeding within 24 hours of the third dose of misoprostol, she should take a fourth dose of misoprostol, included in the study package, as an "extra dose." Instructions for taking other drugs (analgesics, antiemetics and antibiotics), will follow the standard practice of the study provider.

Follow up: A follow-up contact will be scheduled with the participant ten to fifteen days after misoprostol has been administered. The study provider will conduct a telephone interview to assess the abortion outcome. This assessment may include any combination of methods to determine that the client's abortion is complete (patient history, symptom checklist, urine pregnancy test, serum HCG or ultrasound). The study provider will determine together with the participant which option seems most appropriate to her specific situation and will help her find health facilities nearby where they can perform the requested tests, if necessary.

If it is determined that the participant needs an additional dose of misoprostol, she will be instructed to take the additional 4 tablets that were included in the package sent for this purpose provided she did not take them previously due to lack of bleeding. If another dose of misoprostol or other care is required, the participant will be instructed on how and where to obtain it.

Exit interview: When it has been determined that the participant resolved her abortion, she will be asked to complete an exit interview to obtain feedback on the service. The interview is brief and structured and includes questions about her satisfaction with the telemedicine model and whether she had difficulty meeting the requirements.

ELIGIBILITY:
Inclusion Criteria:

* Woman is seeking abortion care and wants to use telemedicine service for her medication abortion procedure.
* Woman has access to an internet connection or a device that allows remote consultation.
* Woman is 15 years of age or older.
* Woman can provide an address to which abortion medications will be mailed.
* Woman reports having no contraindications to a medical abortion.
* The study provider does not suspect ectopic pregnancy or a nonviable pregnancy.
* The gestational age allows sufficient time for the woman to take the misoprostol no later than 84 days of gestation.
* A feasible plan is made that the woman agrees to confirm complete abortion and to seek care to manage incomplete abortion complications.
* The woman understands the study procedures and is likely to comply with study instructions and has granted informed consent to participate in the study.

Exclusion Criteria:

* Medically ineligible for procedure.
* Provider determines that a medical abortion using the telemedicine approach is not appropriate for that person.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events (safety) | 6 weeks
  Incidence of adverse events among those who self-administered medication abortion regimen

SECONDARY OUTCOMES:
Feasibility of telemedicine service | 6 weeks
  Number of reported difficulties related to adhering to requirements of the protocol.
Acceptability of telemedicine service | 6 weeks
  Reported satisfaction levels among participants (very satisfied, satisfied, unsatisfied, very unsatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (3):
- Ecuador (3):
  - El Comité de Derechos Sexuales y Reproductivos de Ecuador (CODESER), Ambato
  - Cemoplaf, Quito
  - Federación Nacional de Obstetrices y Obstetras del Ecuador (FENOE), Quito

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pena M, Figueroa Flores K, Munoz Ponce M, Facio Serafin D, Camarillo Zavala AM, Ruiz Cruz C, Ortiz Salgado IG, Ochoa Rosado Y, Socarras T, Pacheco Lopez A, Bousieguez M. Telemedicine for medical abortion service provision in Mexico: A safety, feasibility, and acceptability study. Contraception. 2022 Oct;114:67-73. doi: 10.1016/j.contraception.2022.06.009. Epub 2022 Jun 24. PMID 35753406
- [Background] Raymond EG, Weaver MA, Shochet T. Effectiveness and safety of misoprostol-only for first-trimester medication abortion: An updated systematic review and meta-analysis. Contraception. 2023 Nov;127:110132. doi: 10.1016/j.contraception.2023.110132. Epub 2023 Jul 29. PMID 37517447
- [Background] Sheldon WR, Durocher J, Dzuba IG, Sayette H, Martin R, Velasco MC, Winikoff B. Early abortion with buccal versus sublingual misoprostol alone: a multicenter, randomized trial. Contraception. 2019 May;99(5):272-277. doi: 10.1016/j.contraception.2019.02.002. Epub 2019 Mar 1. PMID 30831103